CLINICAL TRIAL: NCT02147652
Title: Assessing the Effects of a Personalized Music Therapy With Headphones on Agitation in Patients With Dementia
Brief Title: Personalized Music Therapy and Agitation in Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, MD, FRCPC, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-7490-DE
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease; Vascular Dementia
Keywords: moderate dementia; severe dementia; Alzheimer's disease; Vascular dementia; agitation; personalized music therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Dementia; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Personalized music (Experimental)
  Interventions: Other: Personalized music

INTERVENTIONS:
Other: Personalized music

SUMMARY:
Symptoms of agitation include abuse or aggressive behaviour toward self or others, appropriate behaviour performed with inappropriate frequency, or behaviours that are inappropriate according to social standards. In the later stages of dementia agitation can contribute significantly to patient distress and caregiver stress, and has been associated with poor quality of life. Previous research studies have shown some evidence that personalized music played in daily care situations reduces agitation. The purpose of this study is to evaluate the effects of personalized music therapy via headphones on agitation during hygiene care (grooming).

This study will involve 60 in-patients of the Geriatric Psychiatry ward of Toronto Rehabilitation Institute. The study would take place over the span of 2 weeks and would involve listening to personalized and either non-personalized or no music during daily hygiene care (grooming). Enrolment is completely voluntary and all personal data obtained will remain confidential.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia with possible or probable cause of Alzheimer's disease, Vascular disease, mixed dementia;
* moderate stage of dementia, a score of <20 on MMSE;
* Age 60 to 90 inclusive;
* Preserved hearing (hearing aids are permissible);
* Pittsburgh agitation scale score of ≥ 3 on at least on 3 occasions over a period of 5 days.

Exclusion Criteria:

* auditory deficits requiring correction beyond hearing aids.
* no substitute decision maker available to indicate music preference and patient unable to answer for themselves.
* recent acute event eg. MI, fractures, or major infection (not UTI)
* patients receiving standing orders of medication for personal care

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10-14 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Changes in agitation | 2 weeks
  Changes in agitation as measured by the Pittsburgh agitation questionnaire and "as needed" psychotropic medications for agitation required during hygiene care will be quantitatively assessed. Statistical analyses will be performed to compare levels of agitation and use of "as needed" psychotropic medications for agitation with personalized music therapy with headphones and non-personalized music intervention or usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Tartaglia, MD, FRCPC, Principal Investigator — Assistant Professor, University of Toronto; Toronto Western Hospital, University Health Network; Tanz Centre for Research in Neurodegenerative Disease

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Steen JT, van der Wouden JC, Methley AM, Smaling HJA, Vink AC, Bruinsma MS. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2025 Mar 7;3(3):CD003477. doi: 10.1002/14651858.CD003477.pub5. PMID 40049590